CLINICAL TRIAL: NCT02365155
Title: Effectiveness of an Interdisciplinary Intervention on Frailty Geriatric Patients With Heart Failure.
Brief Title: Training Intervention in Heart Failure and Frail Elderly Population
Acronym: TIHFEP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de la Ribera (Other)
Collaborators: University of Valencia (Other)
Responsible Party: Principal Investigator, Josep Esteve Portalés., Medicine doctor., Hospital de la Ribera
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRibera
Record Dates: First submitted 2015-02-04; First posted 2015-02-18 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Physical Activity
Keywords: Frailty; Heart failure; Physical activity; Cognitive state
MeSH Terms: conditions — Motor Activity; Frailty; Heart Failure | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group. (Experimental): Multicomponent training intervention; Nutrition intervention; Cognitive intervention; D-vitamin intervention; Occupational intervention; Heart failure follow up.
  Interventions: Other: Multicomponent training intervention.; Other: Nutrition intervention; Other: Cognitive intervention; Other: D-vitamin intervention; Other: Occupational intervention; Other: Heart failure follow up.
- Control group. (Active Comparator): Nutrition intervention; Cognitive intervention; D-vitamin intervention; Occupational intervention; Heart failure follow up.
  Interventions: Other: Nutrition intervention; Other: Cognitive intervention; Other: D-vitamin intervention; Other: Occupational intervention; Other: Heart failure follow up.

INTERVENTIONS:
Other: Multicomponent training intervention. — The intervention group will be included in a program specifically developed for this study based on the multidimensional continuous care of patients with heart failure and frailty diagnosis or prefrailty. A joint interdisciplinary nursing intervention including a physical part (endurance, strength, flexibility and balance).
  Arms: Intervention group.
Other: Nutrition intervention — Both groups will be included in a program of quarterly monitoring receiving nutritional support: nutritional advice plus enteral supplementation should specify.
Other: Cognitive intervention — Both groups will be included in a program of quarterly monitoring receiving cognitive support: detection and treatment of depression and delirium in medical consultation.
Other: D-vitamin intervention — Both groups will be included in a program of quarterly monitoring receiving hormonal support: supplementation of vitamin D if required with adjustment for guides.
Other: Occupational intervention — The intervention group will be included in a program specifically developed for this study based on the multidimensional continuous care of patients with heart failure and frailty diagnosis or prefrailty. A joint interdisciplinary nursing intervention including occupational support.
Other: Heart failure follow up. — Both groups will be included in a program specifically developed for this study based on the multidimensional continuous care of patients with heart failure and frailty diagnosis or prefrailty. A joint interdisciplinary medical intervention including and pharmacological treatment of heart failure and comorbidities adjusted according to recent clinical guidelines requirements.

SUMMARY:
There is enough scientific evidence of the benefits detection of frailty in patients with heart failure, which is an important prognostic factor. The usefulness of screening frailty as flattering tool making diagnostic and therapeutic decisions in patients with heart failure and now emerges in various recent studies. However, it is not found in the literature any study on the potential effectiveness of a comprehensive intervention on the fragility that includes the physical section (endurance, strength, flexibility and balance), nutritional, hormonal (supplementation deficit D vitamin) and pharmacological (adjusted to clinical guidelines according to requirements) in patients with heart failure after hospitalization for cardiac decompensation, to improve survival and reduce cardiac decompensation and hospital admissions resulting in a better quality of life for these patients. Therefore, the investigators designed the following study.

DETAILED DESCRIPTION:
HYPOTHESIS Comprehensive intervention fragility in patients older than 70 years after hospitalization for cardiac decompensation improves survival and quality of life of these patients and reduces decompensation and hospital admissions.

OBJECTIVES

Main objective:

1. Check if a comprehensive program of frail elderly patients diagnosed with heart failure improves survival in patients with heart failure.

Secondary objectives:

1. Improving the quality of life and functional parameters of patients with fragility and heart failure.
2. Check if a comprehensive program on the fragility reduces the number of emergency room visits, outpatient specialties involved and hospital admissions.

MATERIAL AND METHODS

Study Design

The investigators have designed a randomized intervention study with control group, unpaired, for a period of up of 12 months.

The intervention group will be included in a program specifically developed for this study based on the multidimensional continuous care of patients with heart failure and frailty diagnosis or prefrailty. A joint interdisciplinary nursing intervention including a physical part (endurance, strength, flexibility and balance), nutrition (enteral nutritional advice plus supplements should specify), cognitive (detection and treatment of depression and delirium in medical consultation) will take, hormonal (Vitamin D supplementation if required to adjust as guides) (Annex 1), occupational and clinical guidelines pharmacological adjusted according to requirements (Annex 1), pre-frail older than 70 years fragile patients over a period of 12 months follow-up after admission for decompensated heart failure, either as primary or secondary diagnosis.

The control group will be included in a program of quarterly monitoring receiving nutritional support (nutritional advice plus enteral supplementation should specify), cognitive (detection and treatment of depression and delirium in medical consultation), hormonal (supplementation of vitamin D if required with adjustment for guides) (Annex 1) and pharmacological treatment of heart failure and comorbidities adjusted according to recent clinical guidelines requirements (Annex 1) in over 70 pre-frail and frail patients over a period of 12 months follow-up after entering for decompensated heart failure, either as primary or secondary diagnosis.

In both groups the initial recruiting visit will take place during hospitalization, attending for inclusion to its pre decompensation leading to admission baseline, using the "CSHA Clinical Frailty Scale" and including patients presenting a score of 4, 5 or 6 in the same (vulnerable, moderate brittleness and fragility light).

Sample The University Hospital of Ribera serves a population of 263,006 inhabitants according to the National Statistics Institute in 2011, of which 13.5% are over 70 years old. Of these, a prevalence of about 15% fragility of prefrailty 34 and 48.8% of 8-17% is estimated cardiaca43 failure. It is estimated that 54% of patients over 70 with heart failure are frail.

Sample size Has increased accuracy of 5%, maintaining a level of confidence of the study in 95%, with an estimated 12 months 5% of the sample and a ratio of estimated loss of 10% mortality in size is obtained sample of 476 individuals in total, divided into two groups: 238 in the intervention group and 238 in the control group.

The recruitment of patients was performed continuously until the required sample size for the study, thus ending it after completing one year of follow the last individual recruited.

SCHEDULE Visit 0. Both groups. During the first 72 hours of hospitalization. Delivery of the patient information leaflet and informed (Annex 3) in the event that consent to be included in the study after previous explanation detailed by physician consent.

-Randomization patient in one of two groups.

VALUATION

* Assessment And comprehensive geriatric nurse.
* Delivery Date next visit within 15 days after discharge with a margin of three days to possible problems of administrative subpoena.
* Making ECG and Rx. thorax.
* Analytical Determination (complete blood count, renal function, liver function, total protein, albumin, C-reactive protein, total cholesterol, fibrinogen, D-dimer, TSH, T4, calcidiol, PTH and iron metabolism. In addition, mining especially for determination of molecular parameters related to oxidation.
* Determination special analytical for determination of molecular parameters related to oxidation. A determination at least 15 days after hospital discharge and at the end of the year will be tracked:

  * Plasma malondialdehyde (High performance liquid chromatography).
  * Plasma oxidized proteins (Western blotting).
  * Serum interleukin (IL) -6 and tumor necrosis factor (TNF) -α (ELISA Kits).
  * Plasma GDF-11 (Western blotting).
  * Plasma Meterorin-like (ELISA Kit).

Will collected a number of epidemiological, anthropometric, clinical and social field with the data obtained in the assessment questioning the patient by the basal state before the onset of clinical deterioration leading to admission variables. These same variables will be used for the assessment of patients in successive visits.

* After hospital discharge, will be made by the attending physician during hospitalization, adjust treatment of heart failure and other comorbidities according to recent clinical guidelines published (Appendix 1).
* Only For the intervention group:
* Explanation to the intervention group plan exercises to do at home, beginning the same from the first visit post-hospitalization.

VISITS AFTER HOSPITALIZATION

* The quarterly medical visits (intervention group and control group) were conducted in the outpatient clinic of Hospital de la Ribera, Alzira (Valencia) by a physician. They must be equipped with computer with SIAS, GAIA and Internet system, and printer, telephone, table and electrocardiograph. The analytical and radiographic controls were carried out by the central service of the same hospital.
* The Monthly visits nursing (only the intervention group) were sent to the address of less coincident with quarterly patient medical examination, to be performed in the outpatient clinic of the Hospital de la Ribera, Alzira (Valencia). These monthly visits will be conducted by a group of nurses available and graduate physiotherapist and educated in heart failure and for physical and functional assessment of patients.
* The Quarterly visits nursing (intervention group and control group) were conducted in the outpatient clinic of Hospital de la Ribera, Alzira (Valencia) coinciding with the quarterly medical assessments. These quarterly visits were also made by a group of nurses available / os and graduate physiotherapist and educated in heart failure and for physical and functional assessment of patients.

He will provide nurses, physiotherapist and optional paper from a notebook with all the variables described in the card 0 and an identification number for each patient after its completion in successive visits, facilitating the collection and storage of confidential data.

INTERVENTION GROUP

* SCHEDULE OF MEDICAL VISITS:
* Visit 1: 15 days after hospital discharge with a lead-time of three days to adjust for possible administrative needs.

  o The current comprehensive geriatric assessment described in the previous section also collected the tests and scales established for this study (Appendix 2) at the time of hospital discharge were performed.
* Visit 2: 3 months after the visit 1, with a timeframe of three days to adjust for possible administrative needs.
* Visit 3: three months after the visit 2, with a timeframe of three days to adjust for possible administrative needs.
* Visit 4: 3 months after the visit 3, with a timeframe of three days to adjust for possible administrative needs.
* Visit 5: 3 months after the visit 4 with a lead-time of three days to adjust for possible administrative needs.

CONTROL GROUP

* SCHEDULE OF MEDICAL VISITS:
* Visit 1: 15 days after hospital discharge with a lead time of three days to adjust for possible administrative needs.

  o The test variables and scales established for this study (Appendix 2) in the present moment and discharge were collected.
* Visit 2: 3 months after the visit 1, with a timeframe of three days to adjust for possible administrative needs.
* Visit 3: three months after the visit 2, with a timeframe of three days to adjust for possible administrative needs.
* Visit 4: 3 months after the visit 3, with a timeframe of three days to adjust for possible administrative needs.
* Visit 5: 3 months after the visit 4 with a lead time of three days to adjust for possible administrative needs.

Statistical treatment

The variables of this study were collected in an Excel table, version 2003 and statistical analysis was performed using the SPSS Windows version 15.0 (SPSS Inc., Chicago, IL).

Categorical variables were described as percentages and continuous variables using the mean value, the standard deviation and confidence interval of 95%. In the bivariate analysis technique Student's t-Fisher to compare means and Pearson Chi-square and linear tendency Mantel-Haenszel for comparison of proportions and the Pearson correlation was used for quantitative variables. Take as the threshold for statistical significance p less than 0.05.

A survival study was performed. The survival will be estimated by the statistical technique of Kaplan-Meier and to determine differences in survival between groups Mantel-Haenszel test was used. Variables associated with mortality at 6 months, using a model of Cox proportional hazards will be studied.

Difficulties and limitations of the study Being a population-based study of over 70 years, the main difficulty recruiting, in addition to performing a comprehensive intervention that includes a portion of physical activity, the investigators have to exclude patients unfit for its baseline for those years . Another difficulty is the need to find nursing staff trained to supervise exercises at home and understanding and significance of rating scales and test for proper completion.

Limitations of the study are that data from the population sample may not apply to other Spanish populations. Another limitation is that only patients with fragility will include established and not prefrágiles, which also could benefit from the program. Failure to have a system of structured communication with primary care physicians and service "ad hoc" emergency for this study, may decrease its effectiveness.

Other Considerations Given the significant number of comorbidities of our patients and multidisciplinary management that entails, will require numerous clinical guidelines for the proper functioning of the study, which is called in this ANNEX text 1 and Annex 2, will be provided to the ethics committee on digital media (USB) towards facilitating its valuation. With regard to informed consent and patient information sheet, be provided in paper and digital format (USB).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 70 years.
2. Individuals hospitalized in internal medicine at the Hospital de la Ribera with primary or secondary diagnosis of heart failure as before:

   I. Clinical heart failure criteria. (Clinical Practice Guidelines 2012 HF) (Annex 1).

   II. Evidence of ventricular systolic or diastolic dysfunction on echocardiographic (TTE).
3. Pre-frailty or frailty according to the Fried frailty scale, fulfilling at least 1 criterion.
4. Signature reported for inclusion in the study consent.

Exclusion Criteria:

1. Expectation of life less than one year.
2. Cancer Patient in active treatment with chemotherapy / biotherapy or radiotherapy.
3. Major surgery within 6 months prior to baseline.
4. Barthel score ≤ 50 points.
5. Moderate to severe cognitive impairment measured by GDS ≥ 5
6. Severe valvular measured by echocardiogram in the last 6 months.
7. Percutaneous or surgical coronary revascularization in the last 3 months.
8. Acute coronary event in the last month.
9. Dyspnoea baseline NYHA IV / IV.
10. COPD / Asthma severe degree or other pathology that conditions severe impairment of lung function.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-06 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Mortality | 365 days (plus or minus 3 days)
  The primary study endpoint is the mortality reduction.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | 365 days(plus or minus 3 days)
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Short Physical Performance Battery and Physical Performance Test | 365 days(plus or minus 3 days)
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Composite effect of a multicomponent training intervention on systemic biomarkers of frailty | 365 days(plus or minus 3 days)
  * Plasma malondialdehyde (High performance liquid chromatography)
  * Plasma oxidized proteins (Western blotting)
  * Serum interleukin (IL)-6 and tumor necrosis factor (TNF)-α (ELISA Kits)
  * Plasma GDF-11 (Western Blotting)
  * Plasma Meterorin-like (ELISA kit)
Geriatric Depression Scale | 365 days(plus or minus 3 days)
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.
Quality of life: EuroQol-5D | 365 days(plus or minus 3 days)
  Change from baseline to the end of the intervention, and the change between the intervention group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco J Tarazona-Santabalbina, MD, PhD, Study Director — Hospital Universitario de la Ribera; Eduardo Rovira Daudi, MD, PhD, Study Director — Hospital Universitario de la Ribera; Carmen Gomez-Cabrera, MD, PhD, Study Director — University of Valencia; Jose Viña Ribes, MD, PhD, Study Director — University of Valencia; Maria Pilar Perez Ros, Nurse, PhD, Study Director — Catholic University of Valencia; Francisco Martínez Arnau, Physio, PhD, Study Director — University of Valencia
Locations (1):
- Hospital Universitario de la Ribera, Alzira, Valencia, Spain